CLINICAL TRIAL: NCT07326553
Title: A Randomized, Open-Label Trial Evaluating the Efficacy of Placental Membrane Dressings in Accelerating Diabetic Foot Healing Compared to Matched Historical Controls Receiving Standard of Care
Brief Title: Efficacy of Placental Membrane Dressings in Accelerating Diabetic Foot Healing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: BioXTek (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX-PM-DW-101
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diabete Mellitus; Foot Ulcer Chronic
MeSH Terms: conditions — Diabetes Mellitus | interventions — membrane-associated placental tissue protein 1

STUDY DESIGN:
Intervention Model Description: Compared to historical controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placental Membrane Dressing (Experimental)
  Interventions: Biological: Placental Membrane
- Historical Controls (No Intervention)

INTERVENTIONS:
Biological: Placental Membrane — Dehyrdated Placental Membrane
  Arms: Placental Membrane Dressing

SUMMARY:
Evaluation of Efficacy of Placental Membrane Dressings in Accelerating Diabetic Foot Healing

ELIGIBILITY:
Inclusion Criteria.

1. Patient has signed the informed consent form.
2. Male or female patient at least 18 years of age or older, as of the date of the screening visit.
3. Confirmed diagnosis of Type 1 or Type 2 DM.
4. Has a DFU that is located below the malleoli ranging in size from 1.0 cm2 to 20.0 cm2, post debridement, when measured by the investigator staff at the screening visit using the eKare device.
5. The DFU has been present for ≥4 weeks and ≤12 months.
6. The DFU is non-healing as defined as <30% reduction in size in response to standard of care from Screening (Visit 1) to Study Day 1 (Visit 2).
7. If more than one ulcer is present the selected target ulcer must be at least 2 cm from the nearest edge of any adjacent ulcers.
8. The depth of the target foot ulcer is graded as Wagner Grade I or II, i.e., with no evidence of exposed muscle, tendon, bone, or joint capsule.
9. Arterial supply adequacy to the foot with the target ulcer confirmed by any one of the following and documented in medical record/EMR:

   1. Great toe pressure ≥ 40 mm/Hg
   2. Systolic blood pressure Ankle Brachial Index (ABI) in the range ≥ 0.70 ≤ 1.20
   3. TcPO2 ≥ 30 mmHg from the foot
   4. Toe Brachial Index or TBI ≥ 0.65
10. Willing to follow all instructions given by the Investigator, return for all visits, and adhere to off-loading protocols while on the study.

Exclusion Criteria

1. Hemoglobin A1c (HbA1c) level is > 10%.
2. Chronic oral steroid use of > 7.5 mg daily within the previous 30 days preceding screening.
3. Chronic oral or parenteral corticosteroids, or any cytotoxic agents within the previous 30 days preceding screening.
4. Has tested positive for Human Immunodeficiency Virus (HIV) or has Acquired Immune Deficiency Syndrome (AIDS).
5. Has malignancy or history of cancer in 5 years preceding the screening visit other than non- melanoma skin cancer.
6. Pregnant or lactating women.
7. Women of child-bearing potential who are unwilling to avoid pregnancy or use an effective form of birth control.
8. Currently on dialysis or planning to start dialysis.
9. Is currently enrolled or participated in another device, drug, or biological trial within 30 days of screening.
10. Has used wound treatments with enzymes, growth factors, living skin, dermal substitutes including other amniotic or umbilical cord tissue therapies, or other advanced biological therapies within the last 30 days.
11. Current use of topical anti-microbial or silver-containing products.
12. Target ulcer is over an active or inactive Charcot deformity.
13. The depth of the target ulcer is graded as Wagner Grade III or higher, i.e., with evidence of exposed muscle, tendon, bone, and/or joint capsule.
14. Gangrene is present on any part of the affected foot.
15. Current suspicion of osteomyelitis, cellulitis, or other clinical signs or symptoms of target ulcer infection.
16. Any previous use of human placental membrane applied to the target ulcer.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks
  Proportion of subjects achieving ≥90% wound closure.

SECONDARY OUTCOMES:
Time to wound closure | 12 weeks
  Time in number of days to ≥90% wound closure over the 12- week treatment period, starting from baseline to the time of initial observation of wound closure
Percent Change | 12 weeks
  Percent change from baseline in wound surface area (cm2)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Axsendo, Phoenix, Arizona
  - Axsendo Clinical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Plan Description De-identified individual participant data (IPD) collected during the study will be made available to qualified researchers. Shared IPD will include participant-level demographic and baseline characteristics, wound characteristics, treatment assignment, and outcome measures related to diabetic foot ulcer healing (e.g., wound closure status, time to closure, wound area measurements, and adverse event data), as well as relevant analyzable datasets. Data will be shared in a de-identified format and will not include direct identifiers.
  Access Criteria Access to de-identified IPD will be provided upon reasonable request to the study sponsor/principal investigator after publication of the primary results. Requests must include a research proposal and statistical analysis plan and will be reviewed for scientific merit and compliance with applicable ethical and privacy requirements. Data will be shared under a data use agreement and may be accessed through a secure data-shar